CLINICAL TRIAL: NCT03554850
Title: Trevo® Retriever Registry (China)
Status: Completed | Type: Observational
Sponsor: Stryker Neurovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: CDM10001400
Record Dates: First submitted 2018-05-23; First posted 2018-06-13 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Real World Data in China

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Trevo® Retriever — Stent retriever procedure

SUMMARY:
Trevo® Retriever Registry (China) is to assess real world performance of the FDA cleared Trevo Retriever intended to restore blood flow in the neurovasculature by removing thrombus in patients experiencing ischemic stroke in China.

DETAILED DESCRIPTION:
Trevo Registry (China) is a prospective, open-label, multi-center study, and it is the first Stryker China trial. This trial assesses real world performance of the Trevo® Retriever which is intended to restore blood flow in the neurovasculature by removing thrombus in subjects experiencing ischemic stroke. Total of 200 subjects among up to 15 sites in China local will participate in this trial. The primary endpoint is revascularization status assessment at the end of the procedure using the modified TICI score.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18
2. Subjects experiencing acute ischemic stroke due to a large vessel occlusion who are eligible and suitable for restoration of blood flow using any approved Trevo Retriever in the neurovasculature to remove thrombus
3. Trevo Retriever is planned to be the primary mechanical neuro-thrombectomy device to remove the thrombus
4. Subject or subject's legally authorized Representative (LAR) has signed the study Informed Consent Form
5. Subject willing to comply with the protocol follow-up requirements

Exclusion Criteria:

1. mRS >2
2. Any known coagulopathy
3. Anticipated life expectancy less than 3 months
4. Known absolute contraindications to the use of required study medications or agents (e.g., heparin, aspirin, clopidogrel, radiographic contrast agents, etc.)
5. Preexisting neurological or psychiatric disease that would prevent complete the study required evaluations
6. The subject is participating in another mechanical neuro-thrombectomy device trial or any other clinical trial where the study procedure or treatment might confound the study end point.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Populations met the inclusion/exclusion criteria above
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2021-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ZhongRong Miao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (10):
- China (10):
  - Beijing TianTan Hospital, Beijing, Beijing Municipality
  - The Hospital of Shunyi District Beijing, Beijing, Beijing Municipality
  - Qingyuan City People's Hospital, Qingyuan, Guangdong
  - The Third Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Puyang Oilfield General Hospital, Puyang, Henan
  - Linyi People's Hospital, Linyi, Shandong
  - Qingdao Central Hospital, Qingdao, Shandong
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Wenzhou Central Hospital, Wenzhou, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrollment occurs when the Trevo Retriever is deployed as the first mechanical neuro-thrombectomy device used to remove the thrombus. A Screening and Enrollment Log will be maintained by each site to document basic information such as date screened and reason for screen failures for subjects who fail to meet the study eligibility criteria. In order to avoid bias, every effort should be made to include all Trevo cases performed over a given duration of time in the registry.
Groups:
- Single Arm-Trevo® Retriever: All subjects who meet the inclusion/exclusion criteria and where Trevo Retriever is used as the initial mechanical thrombectomy device to remove thrombus from the neurovasculature in the setting of acute ischemic stroke.
Period: Overall Study
Arm/Group | Single Arm-Trevo® Retriever
Started | 201
Completed | 190
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Subject Demographics and Baseline Characteristics: Subjects' demographic characteristics will be summarized using descriptive statistic methods.- Continuous variables will be summarized by mean±SD, median, minimum and maximum. Categorical variables will be summarized by percentages and frequencies.
Arm/Group | Subject Demographics and Baseline Characteristics
Number analyzed (Participants) | 201
Age, Categorical [Count of Participants; unit: Participants] — Age will be summarized by percentages and frequencies.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 111
    >=65 years | 90
Age, Continuous [Median (Full Range); unit: years] — Age will be summarized by mean±SD, median, minimum and maximum.
  years | 63 [52 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  China | 201

OUTCOME MEASURES:

1. Primary Outcome: the Modified TICI(Thrombolysis in Cerebral Infarction) Scale at the End of Procedure
Description: The primary endpoint is measured using the modified TICI scale at the end of procedure.Success of primary endpoint was defined as a modified TICI score of 2b or better at the end of procedure. Primary endpoint will be analyzed by percentages, frequencies and the 95% confidence interval of the percentage of success. The 95% confidence interval will be calculated using ClopperPearson exact method.
  Note: Modified TICI score has 6 grades: 0(No Perfusion), 1(Penetration with Minimal Perfusion), 2(Partial Perfusion), 2a(Partial filling with <50% of the entire vascular territory is visualized), 2b(Partial filling with ≥50% of the entire vascular territory is visualized), 3(Complete Perfusion). Higher scores mean a better outcome.
Time Frame: At the end of the neuro-thrombectomy procedure (Day 1)
Population: The Trevo Retriever was used as the primary device in all subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Primary Effectiveness Outcome: post-procedural eTICI score (≥2b)
Arm/Group | Primary Effectiveness Outcome
Number analyzed (Participants) | 190
Participants | 187

2. Secondary Outcome: Day 90 mRS
Description: good clinical outcomes defined as mRS of 0-2.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Groups:
- Day 90 mRS Data: good clinical outcomes defined as mRS of 0-2.
Arm/Group | Day 90 mRS Data
Number analyzed (Participants) | 201
Participants | 148

3. Secondary Outcome: Day 90 Mortality
Description: If the subjects had completed their 90-day visit, the subjects will be considered as alive at Day 90. If the subjects did not come for their Day 90 visit and died, the date of death will be used to compare with the upper window of their Day 90 (90 + 14 days post procedure). If the subjects died after the upper window of their Day 90, the subjects will be considered as alive at their Day 90. Otherwise, the subjects will be counted as death before Day 90.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Groups:
- Day 90 Mortality: If the subjects had completed their 90-day visit, the subjects will be considered as alive at Day 90. If the subjects did not come for their Day 90 visit and died, the date of death will be used to compare with the upper window of their Day 90 (90 + 14 days post procedure). If the subjects died after the upper window of their Day 90, the subjects will be considered as alive at their Day 90. Otherwise, the subjects will be counted as death before Day 90.
Arm/Group | Day 90 Mortality
Number analyzed (Participants) | 201
Participants | 11

4. Secondary Outcome: Neurological Deterioration
Description: Four or more points increase in the NIHSS score from the baseline to 24 hours post procedure.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Groups:
- Neurological Deterioration: Four or more points increase in the NIHSS score from the baseline to 24 hours post procedure.
Arm/Group | Neurological Deterioration
Number analyzed (Participants) | 195
Participants | 15

5. Secondary Outcome: Rate of Study Device and Procedure Related SAE Through Day 90
Description: Rate of study device and procedure related serious adverse events (SAE) through Day 90.
Time Frame: Day 90
Measure: Count of Participants; unit: Participants
Groups:
- Rate of Study Device and Procedure Related SAE Through Day 90.: Rate of study device and procedure related serious adverse events (SAE) through Day 90.
Arm/Group | Rate of Study Device and Procedure Related SAE Through Day 90.
Number analyzed (Participants) | 201
Participants | 0

ADVERSE EVENTS:
Time Frame: If the subjects completed their 90-day visit, the subjects were considered as alive at Day 90. If the subjects did not come for their Day 90 visit and died, the date of death was used to compare with the upper window of their Day 90 (90 + 14 days post procedure). If the subjects died after the upper window of their Day 90, the subjects were considered as alive at their Day 90. Otherwise, the subjects were counted as deaths before Day 90.
Description: The Adverse Events will be monitored/accessed without regard to the specific Adverse Event Term.
Groups:
- Overall Summary of All AEs and SAEs: All SAEs through Day 90 will be summarized by number of events, number of subjects with events and the percentages of subjects with events by the type of SAEs and by their relatedness.
  All AEs during procedure will be summarized by number of events, number of subjects with events and the percentages of the subjects with events by the type of AEs and by their relatedness.
Arm/Group | Overall Summary of All AEs and SAEs
All-Cause Mortality (participants affected / at risk) | 11/201
Serious Adverse Events (participants affected / at risk) | 11/201
Other Adverse Events (participants affected / at risk) | 5/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Summary of All AEs and SAEs (N=201)
Nervous system disorders (Nervous system disorders) | 5
Infections and Infestations (Infections and infestations) | 3
General disorders and administration site conditions (General disorders) | 2
cardiac disorder (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.49% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Summary of All AEs and SAEs (N=201)
Nervous system disorders (Nervous system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/50/NCT03554850/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT03554850/SAP_001.pdf